CLINICAL TRIAL: NCT05715814
Title: A Single Arm, Open Label, Pilot Study to Evaluate the Safety and Efficacy of Once Daily 25mg Empagliflozin in Patients on Peritoneal Dialysis With Residual Kidney Function
Brief Title: meChANisms and sAfety of SGLT2 Inhibition in peRitoneal dialYsis
Acronym: CANARY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Sunita Singh, MD, MSc, FRCPC, Clinician Scientist, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-6198
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Peritoneal Dialysis Complication; End Stage Kidney Disease; Sodium-glucose Co-transporter-2 Inhibitors; Kidney Dysfunction; Residual Kidney Function
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — PO once daily
  Other Names: JARDIANCE

SUMMARY:
The primary aim of this study is to determine the safety and mechanisms of SGLT2 inhibition in individuals on peritoneal dialysis (PD) with residual kidney function (RKF).

DETAILED DESCRIPTION:
The importance of RKF on the survival of patients on PD has been demonstrated in several observational studies. Despite this, there are limited pharmacological interventions available to slow the loss of RKF in these patients. There is an unmet need for novel cardiovascular and kidney protective strategies for patients on renal replacement therapies, including PD.

SGLT2 inhibitors have been shown to have both cardiovascular and kidney protective effects in individuals with kidney disease, with and without diabetes. These benefits have been attributed to diverse mechanisms and kidney benefits have been largely attributed to reductions in intraglomerular pressure at the single nephron level, reversibly lowering GFR in the short-term with long-term benefits. However, the beneficial effects of SGLT2 inhibitors have never been studied in patients on dialysis.

The CANARY study will provide insight into the safety and mechanisms of SGLT2 inhibitors in individuals on dialysis with RKF, with and without type 2 diabetes, over a period of 2 weeks. Demonstrating that protective mechanisms associated with SGLT2 inhibitors are intact in patients on PD with RKF would provide a strong rationale for a larger clinical trial to explore the use of these novel drugs in this unique clinical application. Additionally, our proposed study would provide timely mechanistic data to inform clinical decisions in the context of other large clinical trials such as EMPA-KIDNEY. These findings would help physicians make decisions on leaving patients on SGLT2 inhibitors even beyond end-stage kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent.
* Patients aged ≥18 years on PD with RKF defined as at least 250 cc of urine output per day (assessed via 24-hour urine collection) and a minimum measured GFR of 2 ml/min/1.73m2, as measured at least once in the last 3 months.
* Stable PD prescription, as determined by investigators.
* Stable dose of RAAS blockade if on a medication within this class for the last 30 days.

Exclusion Criteria:

* Type 1 diabetes.
* Recent (in the 30 days prior to screening) acute coronary syndrome or cerebrovascular event.
* PD peritonitis within 30 days of screening.
* History of organ transplant, including pancreas, pancreatic islet cells or kidney transplant.
* Planned surgery/procedures or radiologic investigations requiring contrast during the trial.
* Pregnant, planning to become pregnant, or nursing an infant during the study period
* History of any DKA event
* Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells (e.g., malaria, babesiosis, hemolytic anemia) at screening.
* Women who are pregnant, nursing, or who plan to become pregnant whilst in the trial.
* Alcohol or drug abuse within the 3 months prior to screening that would interfere with trial participation based on Investigator's judgement.
* Use of SGLT2 inhibitor within 30 days prior to screening.
* Intake of an investigational drug in another trial within 30 days prior to screening.
* Patient not able to understand and comply with study requirements, based on Investigator's judgment.
* Any other clinical condition that, based on Investigator's judgement, would jeopardize patient safety during trial participation or would affect the study outcome (e.g. immunocompromised patients, active malignancy, patients who might be at higher risk of developing genital or mycotic infections, patients with chronic viral infections, uncontrolled hypertension, cardiorenal and/or hepatorenal syndrome, severe hepatic impairments etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in measured GFR | Before and 2 weeks after initiation of empagliflozin.
  GFR will be determined from the average of creatinine and urea clearance from a 24-hour urine collection.

SECONDARY OUTCOMES:
Rebound in GFR after Cessation of Therapy | 2 weeks
  A GFR measurement will be performed 2 weeks after cessation of empagliflozin, with the aim of capturing the reversible "rebound" in GFR after cessation of therapy.
Change in ultrafiltration volume | 2 weeks
Change in fraction of glucose remaining in the dialysate | 2 weeks
Change in dialysate/plasma creatinine | 2 weeks
Change in dialysate/plasma urea | 2 weeks
Change in sodium dialysate concentration | 2 weeks
Change in glycated hemoglobin (HbA1c) | 2 weeks
Change in systolic and diastolic blood pressure | 2 weeks
Change in body weight | 2 weeks
Change in body composition (percent body mass, body fat, and muscle mass) | 2 weeks
  Bioimpedence measurements will be taken to study the effects of intervention on body composition.
Change in fractional urine excretion of sodium | 2 weeks
  Urinary analysis will be performed to quantify the amount of sodium excretion.
Change in fractional urine excretion of glucose | 2 weeks
  Urinary analysis will be performed to quantify the amount of glucose excretion.
Change in eGFRβ2-microglobulin | 2 weeks
  Blood sample analysis to assess middle molecule clearance.
Change in degree of albuminuria | 2 weeks
  Urinary analysis will be performed to determine if there has been any change in the severity of albuminuria
Change in BNP (NT-proB-type Natriuretic Peptide) | 2 weeks
Change in markers of neurohumoral activation, erythropoiesis, and inflammation. | 2 weeks
The safety of empaglifllozin use in PD patients with RKF with regard to anuria (<100cc/day), volume depletion, diabetic ketoacidosis, genito-urinary infections, PD peritonitis and death will be evaluated. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sunita KS Singh, MD MSc FRCPC, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided